CLINICAL TRIAL: NCT05008354
Title: Investigation of Pyridoxine Effect on Behavioral Adverse Events of Levetiracetam in Adult Patients With Epilepsy
Brief Title: Effect of Pyridoxine on Behavioral Adverse Events of Levetiracetam
Acronym: EPYLEB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nasim Tabrizi (Other)
Collaborators: Mazandaran University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Nasim Tabrizi, Associate professor of neurology, Mazandaran University of Medical Sciences
Organization: Mazandaran University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5238
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Epilepsy; Pyridoxine; Behavior Problem
MeSH Terms: conditions — Epilepsy; Mental Disorders | interventions — Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyridoxine (Active Comparator)
  Interventions: Drug: Pyridoxine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridoxine — Pyridoxine tablet 40mg once daily
  Arms: Pyridoxine
Drug: Placebo — Placebo tablet once daily
  Arms: Placebo

SUMMARY:
This study is a two-arm parallel group randomized double-blind placebo-controlled trial with the aim of Investigating pyridoxine effect on behavioral side effects of levetiracetam in adult patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Patients with epilepsy
* Patients who are treated by levetiracetam (Levebel, Cobel darou) in recent month
* Complaint of behavioral problem
* Patient's consent for participation

Exclusion Criteria:

* History of known psychiatric disease
* Pregnancy
* Incidence of psychotic side effects including hallucination, psychosis, suicidal idea or attempt
* Treatment with psychiatric medications
* Alcohol or drug abuse
* Mental retardation to the degree that intervenes comprehension and response to questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Behavioral side effects | 3 weeks
  Behavioral side effects are measured by SCL-90-R questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Bu Ali Sina Hospital, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: No